CLINICAL TRIAL: NCT00189124
Title: Does DHEA Improve Endothelial Dysfunction and Other Cardiovascular Risk Factors in Premenopausal Women With Systemic Lupus?
Brief Title: Dehydroepiandrosterone (DHEA) in Systemic Lupus Erythematosus (SLE) for Coronary Artery Disease (CAD) Prevention
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Wendy Marder, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2001-0822
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Dehydroepiandrosterone (DHEA); DHEA; SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Dehydroepiandrosterone (DHEA)

SUMMARY:
The purpose of this study is to evaluate the effect of DHEA on endothelial dysfunction in patients with systemic lupus by measuring:

1. changes in brachial artery flow-mediated dilatation (FMD) and
2. changes in biomarkers of cardiovascular risk. Patients will be enrolled in a randomized, double-blinded crossover trial of DHEA or placebo for ten weeks, then crossed over to the alternate treatment arm after a six-week washout period.

HYPOTHESIS: Dehydroepiandrosterone (DHEA) administration in premenopausal women with SLE modifies cardiovascular risk by improving vascular endothelial function and other biomarkers associated with cardiovascular heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Member of the Michigan Lupus Cohort
* Meet the American College of Rheumatology (ACR) criteria for SLE
* Premenopausal

Exclusion Criteria:

* Smoker
* Diabetic
* Prednisone dose > 10 mg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-09; Primary Completion 2005-12 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Brachial artery reactivity, by flow mediated dilatation

SECONDARY OUTCOMES:
Changes in biomarkers of SLE
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Marder, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States